CLINICAL TRIAL: NCT04044989
Title: Placebo-Controlled, Randomized, Double Blind Trial of Effect of Photobiomodulation Therapies On The Root Resorption Associated With Orthodontic Forces: A Pilot Study Using Micro Computed Tomography
Brief Title: Photobiomodulation and Root Resorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Merve Goymen, Asisst. Prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 332
Record Dates: First submitted 2019-07-29; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Orthodontic Pathological Resorption of External Root; Orthodontic Appliance Complication; Orthodontic Tooth Movement
Keywords: photobiomodulation; laser; LED; resorption; micro-CT
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root resorption (total) (Experimental): The resorption cavities on the root surface were determined and the volumes of the cavities were measured in CTAn software (micro-CT).
  Interventions: Device: Laser; Device: light-emitting diode (LED); Device: Placebo
- Root resorption (local) (Experimental): The resorption cavities on the root surface (palatal, buccal, distal and mesial root surfaces) were determined and the volumes of the cavities were measured in CTAn software (micro-CT).
  Interventions: Device: Laser; Device: light-emitting diode (LED); Device: Placebo

INTERVENTIONS:
Device: Laser — Diode laser device was used for photobiomodulation
Device: light-emitting diode (LED) — LED device was used for photobiomodulation
Device: Placebo — Diode laser device was used for placebo effect

SUMMARY:
Objectives: The aim of this study is to investigate the effect of photobiomodulation therapies on root resorption compared with the placebo group. Materials and Methods: 30 patients, who were admitted to the …………. University Faculty of Dentistry Orthodontics Department for treatment, with an indication of upper right 1st premolar tooth extraction was included. Before the individuals' orthodontic treatment, 0.022 slot MBT brackets and tubes were placed on the maxillary 1st premolar and molar. A 150g buccal tipping force was applied to the 1st premolar. Individuals were then randomly divided into 3 groups. For the first group; laser application was performed with a 810 nm GaAlAs laser device at 0,3,7,14,21 and 28 days to 8 J/cm2. Second group; an LED application according to the manufacturer's instructions with a 850 nm wavelength and 20 mW/cm2 output power for 10 minutes per day during the experiment. Third group; a placebo therapy was completed whereby a laser device that did not make active pulses was used. At the end of four weeks, the amount of root surface resorption was compared using micro-CT imaging after the extraction of the teeth.

ELIGIBILITY:
Inclusion Criteria:

* No history of orthodontic treatment
* No systemic disease or craniofacial anomaly
* No dental trauma and tooth with root resorption
* Having good oral hygiene
* No periodontal disease (no more than 3mm pocket)
* No restored or endodontically untreated upper right 1st premolar teeth
* Having the maxillary right 1st premolar tooth extraction indication of orthodontic treatment

Exclusion Criteria:

* Problems in patient compliance
* Inadequate oral hygiene
* Development of any medical problem making orthodontic treatment contraindicated during the study period

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Root Resorption | through study completion, an average of 4 weeks
  Crater volume measurement

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gulec, PhD, Principal Investigator — Gaziantep University Orthodontics Department; Merve Goymen, PhD, Study Chair — Gaziantep University Orthodontics Department
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No